CLINICAL TRIAL: NCT06847659
Title: Comparison of the Effect of Prewarming on Intraoperative Hypothermia in Patients Undergoing HoLEP (Holmium Laser Prostatectomy) Surgery
Brief Title: Comparison of the Effect of Prewarming on Intraoperative Hypothermia in Patients Undergoing Holmium Laser Prostatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Betül Güven, Ankara City Hospital Bilkent, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TABED1-24-841
Record Dates: First submitted 2025-02-18; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Prewarming; Holmium Laser Prostate Surgery; Hypothermia Following Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prewarming Group (Experimental): Patients will receive 10 minutes of 43°C forced-air warming and 41°C prewarmed intravenous fluid before surgery. Surgery will begin following the standard induction of general anesthesia once patients are in the operating room. An air blower set to 43°C will maintain patient warmth throughout the procedure.
  Interventions: Diagnostic Test: intraoperative body temperature
- Control Group (Other): No prewarming will be applied. Surgery will begin following the standard induction of general anesthesia once patients are in the operating room. An air blower set to 43°C will maintain patient warmth throughout the procedure.
  Interventions: Diagnostic Test: intraoperative body temperature

INTERVENTIONS:
Diagnostic Test: intraoperative body temperature — Body temperature measurement with esophageal probe

SUMMARY:
This study aims to evaluate the effectiveness of prewarming methods in preventing intraoperative hypothermia in patients undergoing HoLEP surgery. Designed as a randomized controlled study, patients who receive prewarming will be compared with those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years and older
* Patients undergoing HoLEP surgery under general anesthesia
* Patients who consent to participate in the study

Exclusion Criteria:

* Patients who refuse to participate in the study.
* Patients unable to read, understand, or sign the informed consent form.
* Hemodynamically unstable patients.
* Patients with a preoperative or intraoperative body temperature >37°C.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to onset of intraoperative hypothermia. | intraoperatively
  Time to develop intraoperative hypothermia (when body temperature drops below 36°C)

SECONDARY OUTCOMES:
Hemodynamic parameters | intraoperatively
  heart rate
Volume of irrigation fluid used | intraoperatively
  Volume of irrigation fluid used
Changes in body temperature | intraoperatively
  Changes in preoperative and intraoperative body temperature
Hemodynamic parameters | intraoperatively
  mean arterial pressure
respiratory parameter | intraoperatively
  SpO2

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided